CLINICAL TRIAL: NCT01812330
Title: The Effect of Ticagrelor on Acute Coronary Syndrome Patients With Clopidogrel Resistance Undergoing Percutaneous Coronary Intervention
Brief Title: Efficacy and Safety Study of Ticagrelor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130118 CR
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-03

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; CR; PCI; Platelet funtion; Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Experimental): Group 1 will be administered with Clopidogrel 75mg daily until the end of the trial
  Interventions: Drug: Clopidogrel
- group 2 (Experimental): Group 2 will be administered with Clopidogrel 150mg daily until the end of trial
  Interventions: Drug: Clopidogrel
- group 3 (Experimental): Group 3 will be administered with Ticagrelor 90mg twice daily until the end of the trial
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — After 600mg loading dose, 75mg or 150mg Qd
  Other Names: Plavix
  Arms: group 1; group 2
Drug: Ticagrelor — 90mg Bid
  Other Names: Brilique
  Arms: group 3

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ticagrelor with clopidogrel

DETAILED DESCRIPTION:
180 elective percutaneous coronary intervention patients with clopidogrel resistance were randomized to three groups, Group 1:received clopidogrel 75mg qd ;Group 2:received clopidogrel 150mg qd ; Group 3:received ticagrelor 90mg bid after PCI.Platelet funtion were tested by flowcytometric vasodilator-stimulated phosphoprotein(VASP) analysis before PCI,and 3days,7days and 1 month after PCI,respectively.The aim of our study is to compare the efficacy and safety of ticagrelor with clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of ACS 2.undergoing PCI 3.with clopidogrel resistance

Exclusion Criteria:

* 1.any contraindication against the use of clopidogrel and ticagrel 2.Contradiction to aspirin and contrast medium 3.Life expectancy less than 1 year 4.Tumor or inflammatory diseases5. fibrinolytic therapy within 24 hours before randomization 6.a need for oral anticoagulation therapy 7. an increased risk of bradycardia 8.concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer 9.a history of asthma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
PRI | post operative 1 month
  Platelet funtion were tested by flowcytometric vasodilator-stimulated phosphoprotein(VASP) analysis.And a platelet reactivity index (PRI) was calculated.

SECONDARY OUTCOMES:
Major adverse cardiac events(MACEs) | follow-up for 1 month
  cardiovascular death,angiographically conﬁrmed stent thrombosis, recurrent acute coronary syndrome deﬁned by the American College of Cardiology/American Heart Association guidelines,and recurrent revascularization by either coronary angioplasty or bypass surgery
major and minor bleeding | follow-up for 1 month
  Major bleeding was deﬁned as intracranial bleeding or clinically-overt bleeding associated with a decrease in hemoglobin of 50 g/L, according to the Thrombolysis inMyocardial Infarction (TIMI) criteria .Minor bleeding was also deﬁned according to TIMI criteria .

CONTACTS AND LOCATIONS:
Overall Officials: huiliang liu, doctor, Principal Investigator — Department of Cardiology of General Hospital of Chinese People's Armed Police Forces
Locations (1):
- General Hospital of Chinese People's Armed Police Forces, Beijing, China

REFERENCES:
- [Result] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878
- [Result] Cuisset T, Frere C, Quilici J, Poyet R, Gaborit B, Bali L, Brissy O, Morange PE, Alessi MC, Bonnet JL. Comparison of omeprazole and pantoprazole influence on a high 150-mg clopidogrel maintenance dose the PACA (Proton Pump Inhibitors And Clopidogrel Association) prospective randomized study. J Am Coll Cardiol. 2009 Sep 22;54(13):1149-53. doi: 10.1016/j.jacc.2009.05.050. PMID 19761935
- [Result] Gurbel PA, Bliden KP, Zaman KA, Yoho JA, Hayes KM, Tantry US. Clopidogrel loading with eptifibatide to arrest the reactivity of platelets: results of the Clopidogrel Loading With Eptifibatide to Arrest the Reactivity of Platelets (CLEAR PLATELETS) study. Circulation. 2005 Mar 8;111(9):1153-9. doi: 10.1161/01.CIR.0000157138.02645.11. Epub 2005 Feb 28. PMID 15738352
- [Result] von Beckerath N, Taubert D, Pogatsa-Murray G, Schomig E, Kastrati A, Schomig A. Absorption, metabolization, and antiplatelet effects of 300-, 600-, and 900-mg loading doses of clopidogrel: results of the ISAR-CHOICE (Intracoronary Stenting and Antithrombotic Regimen: Choose Between 3 High Oral Doses for Immediate Clopidogrel Effect) Trial. Circulation. 2005 Nov 8;112(19):2946-50. doi: 10.1161/CIRCULATIONAHA.105.559088. Epub 2005 Oct 31. PMID 16260639
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Jeong YH, Lee SW, Choi BR, Kim IS, Seo MK, Kwak CH, Hwang JY, Park SW. Randomized comparison of adjunctive cilostazol versus high maintenance dose clopidogrel in patients with high post-treatment platelet reactivity: results of the ACCEL-RESISTANCE (Adjunctive Cilostazol Versus High Maintenance Dose Clopidogrel in Patients With Clopidogrel Resistance) randomized study. J Am Coll Cardiol. 2009 Mar 31;53(13):1101-9. doi: 10.1016/j.jacc.2008.12.025. PMID 19324253